CLINICAL TRIAL: NCT05503576
Title: Effect of Mobile Application Usage on Drug Compliance After Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Pinar Kaya, PhD student, Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17992086462
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Drug Compliance; Patient Acceptance of Health Care
Keywords: Thyroidectomy; Nurse; Medication Compliance; Reminder; mobile; application
MeSH Terms: conditions — Medication Adherence; Patient Acceptance of Health Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reminder mobile application group (Experimental): The mobile application will be introduced with a video demonstration. Then, with the help of the researcher, the mobile application will be downloaded to his phone. A user name and password will be created for the patient to enter the application. It will be explained that medication and appointment reminders are available in the application. It will be emphasized that the application will direct you to the hospital appointment system to create a control appointment. In addition, it will be announced that the training content prepared with the contribution of experts to increase drug compliance can be accessed through the application. It is thought that the patient will be interviewed for approximately 20 minutes for the information and procedure process. In the next process, the "Drug Protocol Information Form", "Modified Morisky Scale" and "Complications Follow-up Form" sent to the patient through the application will be filled in at the 1st, 4th, 8th and 12th weeks.
  Interventions: Device: reminder mobile application
- standard protocol group (No Intervention): If the patient is in the control group in group assignment; After the first encounter and obtaining consent, the "Personal Information Form" will be filled in. Next 1., 4.,8. And in the 12th weeks, the "Drug Protocol Information Form", "Modified Morisky Scale" and "Complications Follow-up Form" will be filled in by telephone interviewing the patient. It is estimated that each phone call with the patient for data collection will take approximately 10 minutes.

INTERVENTIONS:
Device: reminder mobile application — After thyroidectomy, patients will be reminded of medication and control appointments. In addition, patients will be able to access up-to-date and short trainings.
  Arms: reminder mobile application group

SUMMARY:
In patients who have undergone thyroidectomy surgery, drug use will be reminded with a mobile application in the postoperative period.

DETAILED DESCRIPTION:
Summary: Thyroidectomy is frequently used in the treatment of multinodular goiter, graves' disease, multinodular toxic goiter, and thyroid malignancies in general surgery practice. The thyroid gland plays an important role in the rate of metabolism. As a result of removal of the thyroid gland, patients may experience hormonal problems. In thyroidectomy patients, hypothyroidism develops directly due to removal of the thyroid gland; Complications due to parathyroid gland damage, such as hypocalcemia, may also be encountered.

In the management of complications in the postoperative period, monitoring of thyroid hormone and calcium levels is of vital importance in patients. In the case of calcium deficiency in patients, calcium replacement is performed. Levothyroxine replacement is applied to correct thyroid hormone deficiency. When the optimal dose of levothyroxine is adjusted and used appropriately, the rate of side effects is very low. Although the appropriate dose for the patients is determined in the process, thyroid hormone stabilization has the potential to deteriorate over the years.

Medication incompatibility is an important problem in thyroidectomy patients who need to receive levothyroxine replacement throughout their lives. Many studies evaluating drug compliance in the literature have been conducted with samples of internal medicine patients. However, drug compliance after thyroidectomy is an acute and important condition. There is a need for interventions to increase drug compliance in this patient group.

Today, mobile applications are becoming a new trend among technological approaches that increase the patient and nurse contact. However, no study has been found in the literature examining the use of mobile applications and drug compliance and drug level monitoring in thyroidectomy patients. In our randomized controlled study, data will be collected from two patient groups, the experimental and control groups, and the effectiveness of the reminder mobile application will be evaluated. While no additional intervention was applied to the patients in the control group; Patients in the experimental group will be provided to use the Reminder Mobile Application. At the end of the study, it is predicted that the Reminder Mobile Application will increase drug compliance and complication management of patients after thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* Having thyroidectomy due to benign thyroids,
* Being between the ages of 18-65,
* Mental status problem,
* Psychiatric experimentation that reduces understanding and communication,
* Hearing and visual impairment,
* Being able to speak, read, read Turkish,
* Total thyroidectomy performed by the same surgeon, and
* Smart android system phone replacement.

Exclusion Criteria:

Patients who do not meet the inclusion criteria in the sample, patients who meet the inclusion criteria but cannot use mobile applications, do not have internet access, and patients who do not approve to participate in the study will be excluded from the study.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
medication compliance | 0-12 weeks
  Thyroidectomy summative mobile application Modified Morisky Scale total score. The scale consists of 6 items in total. Scale questions are answered as Yes/No. In the evaluation, yes is scored as 1 and no as 0 in questions 2 and 5. In other questions, yes is scored 0, no 1. If the total score of the patient in questions 1, 2 and 6 is 0 or 1, it indicates a low motivation level in terms of drug compliance. A score of 2 or above indicates a high motivation level in terms of drug compliance. If the total score obtained from questions 3, 4 and 5 is 0 or 1, it indicates a low level of knowledge about drug compliance. A score of 2 or more indicates a high level of knowledge about drug compliance.